CLINICAL TRIAL: NCT07020988
Title: An Open Label, Single Dose, Randomized, Active Comparator, Quantitative Electroencephalogram Crossover Study to Assess the Time to Onset of Action of Staccato Alprazolam Versus Intravenous Midazolam and of Staccato Alprazolam Versus Nasal Diazepam in Healthy Study Participants
Brief Title: A Study to Assess the Time to Onset of Action of Staccato Alprazolam Versus Midazolam and Diazepam in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP0127
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
Keywords: Phase 1; Staccato alprazolam; midazolam; diazepam; Healthy Study Participants
MeSH Terms: interventions — Midazolam; Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pilot Part (Experimental): Study participants who successfully completed the Screening Period will receive single dose of Intravenous (IV) midazolam on Day 1 of the Intervention Period.
  Interventions: Drug: Midazolam
- Main Part-Group 1: Treatment Sequence AB (Experimental): Study participants randomized in Group 1 will receive Treatment A: Staccato Alprazolam on Day 1 of the Intervention Period 1 followed by Treatment B: IV Midazolam on Day 1 of the Intervention Period 2.
  Interventions: Drug: Staccato Alprazolam; Drug: Midazolam
- Main Part-Group 1: Treatment Sequence BA (Experimental): Study participants randomized in Group 1 will receive Treatment B: IV Midazolam on Day 1 of the Intervention Period 1 followed by Treatment A: Staccato Alprazolam on Day 1 of the Intervention Period 2.
  Interventions: Drug: Staccato Alprazolam; Drug: Midazolam
- Main Part-Group 2: Treatment Sequence AC (Experimental): Study participants randomized in Group 2 will receive Treatment A: Staccato Alprazolam on Day 1 of the Intervention Period 1 followed by Treatment C: Nasal Diazepam on Day 1 of the Intervention Period 2.
  Interventions: Drug: Staccato Alprazolam; Drug: Diazepam
- Main Part-Group 2: Treatment Sequence CA (Experimental): Study participants randomized in Group 2 will receive Treatment C: Nasal Diazepam on Day 1 of the Intervention Period 1 followed by Treatment A: Staccato Alprazolam on Day 1 of the Intervention Period 2.
  Interventions: Drug: Staccato Alprazolam; Drug: Diazepam

INTERVENTIONS:
Drug: Staccato Alprazolam — Study participants will receive single dose of Staccato Alprazolam at pre-specified time points.
  Other Names: UCB7538
  Arms: Main Part-Group 1: Treatment Sequence AB; Main Part-Group 1: Treatment Sequence BA; Main Part-Group 2: Treatment Sequence AC; Main Part-Group 2: Treatment Sequence CA
Drug: Midazolam — Study participants will receive single dose of IV Midazolam at pre-specified time points.
  Arms: Main Part-Group 1: Treatment Sequence AB; Main Part-Group 1: Treatment Sequence BA; Pilot Part
Drug: Diazepam — Study participants will receive single dose of Nasal Diazepam by inhalation at pre-specified time points.
  Arms: Main Part-Group 2: Treatment Sequence AC; Main Part-Group 2: Treatment Sequence CA

SUMMARY:
The purpose of this study is to estimate the difference in the time to onset of action between Staccato alprazolam and intravenous (iv) midazolam using changes in power in the combined spindle and β1 frequency bands in the qEEG (quantitative electroencephalogram).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 20 years to 55 years of age, inclusive, at the time of signing the ICF.
* Participant is overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring, at the Screening Visit and on Day -1 of the single Intervention Period for the Pilot Part or on Day -1 of the first Intervention Period for the Main Part of the study.
* Participant has a bodyweight of at least 45 kilograms (kg) (female) and 50 kg (male) and a body mass index within the range of 18 Kilograms per meter square (Kg/m2) to 30 kg/m2 (inclusive)
* Participant has given informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in protocol.

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the participant's ability to participate in this study.
* Participant has a history of chronic alcohol or drug abuse, as defined in the most recent version of the Diagnostic and Statistical Manual of Mental Disorders, within 6 months prior to the Screening Visit.
* Participant has a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, cerebrovascular, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Participant has a history of or has been diagnosed with epilepsy or epileptic seizures.
* Participant has abnormal EEG findings at Screening including background slowing (<8Hz), focal slowing (focal δ-activity), or epileptiform discharges.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Time to reach a z-score of absolute power >2 and maintained for at least 60 seconds in the combined spindle and β1 frequency bands within the first 60 minutes of study intervention administration of Staccato alprazolam in Group 1 | Within the first 60 minutes of the study intervention administration on Day 1 of the Intervention Period in Group 1
  Time to reach a z-score of absolute power >2 is derived from the z-scores over time for the combined spindle and β1 frequency bands. The z-scores are calculated using an algorithm applied to the quantitative electroencephalogram (qEEG) data recorded for each study participant.
Time to reach a z-score of absolute power >2 and maintained for at least 60 seconds in the combined spindle and β1 frequency bands within the first 60 minutes of study intervention administration of iv midazolam in Group 1 | Within the first 60 minutes of the study intervention administration on Day 1 of the Intervention Period in Group 1
  Time to reach a z-score of absolute power >2 is derived from the z-scores over time for the combined spindle and β1 frequency bands. The z-scores are calculated using an algorithm applied to the quantitative electroencephalogram (qEEG) data recorded for each study participant.

SECONDARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events (TEAEs) from the first study intervention administration to the Safety Follow-Up (SFU) Visit/ Early Termination Visit (ETV) | From the first study intervention administration to the Safety Follow-Up (SFU) Visit/ Early Termination Visit (ETV) (up to 55 Days)
  Treatment Emergent Adverse Events (TEAEs) are any untoward medical incidence in a participant after the administration of study treatment, whether or not these events are related to study treatment.
Occurrence of Serious TEAEs from the first study intervention administration to the Safety Follow-Up (SFU) Visit/ Early Termination Visit (ETV) | From the first study intervention administration to the Safety Follow-Up (SFU) Visit/ Early Termination Visit (ETV) (up to 55 Days)
  Serious Treatment-Emergent Adverse Events (Serious TEAEs) are any untoward medical incidence in a participant during administered study treatment, whether or not these events are related to study treatment and additionally are emergent untoward medical occurrence that at any dose:
  Results in death; Is life-threatening; Requires in patient hospitalisation or prolongation of existing hospitalisation; Results in persistent disability/incapacity; Is a congenital anomaly or birth defect; Important medical events.
Time to reach a z-score of absolute power >2 and maintained for at least 60 seconds in the combined spindle and β1 frequency bands within the first 60 Minutes of study intervention administration of Staccato alprazolam in Group 2 | Within the first 60 minutes of the study intervention administration on Day 1 of the Intervention Period in Group 2
  Time to reach a z-score of absolute power >2 is derived from the z-scores over time for the combined spindle and β1 frequency bands. The z-scores are calculated using an algorithm applied to the qEEG data recorded for each study participant.
Time to reach a z-score of absolute power >2 and maintained for at least 60 seconds in the combined spindle and β1 frequency bands within the first 60 Minutes of study intervention administration of nasal diazepam in Group 2 | Within the first 60 minutes of the study intervention administration on Day 1 of the Intervention Period in Group 2
  Time to reach a z-score of absolute power >2 is derived from the z-scores over time for the combined spindle and β1 frequency bands. The z-scores are calculated using an algorithm applied to the qEEG data recorded for each study participant.
Maximum concentration (Cmax) of alprazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  Cmax=maximum concentration
Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC[0-t]) of alprazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC(0-t)=area under the concentration-time curve from time 0 to the last quantifiable concentration
Area Under the Concentration Time Curve From Time 0 to Infinity (AUC) of alprazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC=area under the concentration-time curve from time 0 to infinity
Maximum concentration (Cmax) of midazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  Cmax=maximum concentration
Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC[0-t]) of midazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC(0-t)=area under the concentration-time curve from time 0 to the last quantifiable concentration
Area Under the Concentration Time Curve From Time 0 to Infinity (AUC) of midazolam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC=area under the concentration-time curve from time 0 to infinity
Maximum concentration (Cmax) of diazepam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  Cmax=maximum concentration
Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC[0-t]) of diazepam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC(0-t)=area under the concentration-time curve from time 0 to the last quantifiable concentration
Area Under the Concentration Time Curve From Time 0 to Infinity (AUC) of diazepam | Plasma samples will be collected at predose (Day 1) and at pre-defined time points upto 24 hours postdose
  AUC=area under the concentration-time curve from time 0 to infinity

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- Up0127 1001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual patient-level data (IPD) cannot be adequately anonymized as, there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.